CLINICAL TRIAL: NCT02654353
Title: A New Approach to Target the Substrates of Persistent Atrial Fibrillation: The Sequential Substrate Ablation Approach
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Thomas Rostock, Prof. Dr. Thomas Rostock, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PersAF-Abl2014
Record Dates: First submitted 2016-01-09; First posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Persistent atrial fibrillation, catheter ablation, outcome
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: stepwise ablation (Other): Stepwise ablation of persistent atrial fibrillation (conventional treatment arm) In this arm, patients will be treated with the conventional stepwiese ablation approach
  Interventions: Procedure: Ablation
- Group B: sequential substrate ablation (Active Comparator): Sequential substrate ablation of persistent atrial fibrillation (novel procedure) In this arm, patients will undergo an ablation procedure that consist of PVI, cardioversion, linear ablation and atrial fibrillation re-induction after blocked lines, followed by electrogram-guided ablation
  Interventions: Procedure: Ablation

INTERVENTIONS:
Procedure: Ablation — In both arms, patients will undergo an ablation procedure for persistent atrial fibrillation. The sequence of ablation steps are different between both arms.

SUMMARY:
This is a prospective randomized controlled trial that compares the conventional stepwise approach with a new sequential substrate ablation approach for persistent atrial fibrillation.

DETAILED DESCRIPTION:
A total number of 100 patients with persistent AF were randomized to receive either conventional stepwise ablation (conventional group) or a sequential substrate ablation (substrate group), both with the endpoint of AF termination. All patients were in AF before the procedure. The sequential substrate ablation consisted of pulmonary vein isolation (PVI) followed by cardioversion and linear ablation at the mitral isthmus, left atrial roof and cavotricuspid isthmus in order to modify the AF substrate. After achievement of bidirectional block, AF was re-induced and electrogram-based ablation was performed to achieve AF termination to sinus rhythm (SR). Endpoints are single-procedure outcome and total amount of RF ablation time required to terminate AF by electrogram-guided ablation.

ELIGIBILITY:
Inclusion Criteria:

* persistent atrial fibrillation lasting longer than 3 months
* no previous ablations
* at least 1 electrical cardioversion

Exclusion Criteria:

* non-persistent atrial fibrillation
* previous ablation procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of patients without any arrhythmias during follow-up of 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rostock, MD, Principal Investigator — University Hospital Mainz, Department of Cardiology
Locations (1):
- University Hospital Mainz, Department of Medicine II, Mainz, Germany